CLINICAL TRIAL: NCT05024032
Title: Efficacy and Safety of Tirzepatide Once Weekly in Chinese Participants Without Type 2 Diabetes Who Have Obesity or Are Overweight With Weight-Related Comorbidities: A Randomized, Double-Blind, Placebo-Controlled Trial (SURMOUNT-CN)
Brief Title: A Study of Tirzepatide (LY3298176) in Chinese Participants Without Type 2 Diabetes Who Have Obesity or Overweight (SURMOUNT-CN)
Acronym: SURMOUNT-CN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17507; I8F-MC-GPIA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-08-25; First posted 2021-08-27 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Overweight; Metabolism and Nutrition Disorder
MeSH Terms: conditions — Obesity; Overweight; Nutrition Disorders | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 10 Milligrams (mg) Tirzepatide (Experimental): Participants received maintenance dose 10 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg, and then 10 mg tirzepatide administered subcutaneously (SC) once weekly (QW).
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received maintenance dose 15 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg and then 15 mg tirzepatide administered SC QW.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received matching placebo SC QW.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 Milligrams (mg) Tirzepatide; 15 mg Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study of tirzepatide in Chinese participants without Type 2 Diabetes who have obesity or overweight.

The main purpose is to learn more about how tirzepatide affects body weight.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI ≥28 kilogram/square meter (kg/m²), or ≥24 kg/m² and previous diagnosis with at least one of the following comorbidities: hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease
* Have a history of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* Have Diabetes Mellitus
* Have a self-reported change in body weight >5 kg within 3 months prior to screening
* Have obesity induced by other endocrinological disorders
* Have had a history of chronic or acute pancreatitis
* Have a history of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Have any lifetime history of a suicide attempt
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- China (29):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhujiang Hospital, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Qingpu Branch of Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The Fifth People's Hospital of Shanghai, Shanghai
  - Shanghai Minhang District Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Zhao L, Cheng Z, Lu Y, Liu M, Chen H, Zhang M, Wang R, Yuan Y, Li X. Tirzepatide for Weight Reduction in Chinese Adults With Obesity: The SURMOUNT-CN Randomized Clinical Trial. JAMA. 2024 Aug 20;332(7):551-560. doi: 10.1001/jama.2024.9217. PMID 38819983

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 Milligrams (mg) Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 70 | 71 | 69
Received At Least One Dose | 70 | 71 | 69
Completed | 69 | 67 | 65
Not Completed | 1 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Deviation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 10 mg Tirzepatide: Participants received maintenance dose 10 mg with dose escalation starting from 2.5 mg, 5 mg, 7.5 mg, and then 10 mg tirzepatide administered SC QW.
- Total: Total of all reporting groups
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 70 | 71 | 69 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.70 (7.24) | 35.80 (9.33) | 37.80 (10.24) | 36.10 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 33 | 103
  Male | 35 | 36 | 36 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 70 | 71 | 69 | 210
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 70 | 71 | 69 | 210
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 92.2 (16.2) | 91.3 (16.2) | 92.0 (15.8) | 91.8 (16.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Body Weight
Description: Mean Percent Change from Baseline in Body Weight. Least squares (LS) mean was determined using mixed model repeated measures (MMRM) model with Baseline + Sex + Presence of Comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
Percent change | -14.4 (0.98) | -19.9 (1.01) | -2.4 (1.00)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.0, 95% CI 2-sided [-14.8 to -9.3]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -17.5, 95% CI 2-sided [-20.3 to -14.8]

2. Primary Outcome: Percentage of Participants Who Achieve ≥5% Body Weight Reduction
Description: Percentage of Participants who Achieve ≥5% Body Weight Reduction. A logistic regression model was used for this analysis.
Time Frame: Week 52
Population: All participants who received at least one dose of study drug and had evaluable body weight data.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
Percentage of participants | 91.43 | 92.65 | 29.41
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 23.11, 95% CI 2-sided [8.80 to 60.69]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 26.53, 95% CI 2-sided [9.61 to 73.24]

3. Secondary Outcome: Mean Change From Baseline in Body Weight
Description: Mean Change from Baseline in Body Weight. LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 20
Population: All participants who received at least one dose of study drug and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
kilograms (kg) | -9.0 (0.59) | -11.1 (0.61) | -1.8 (0.60)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.2, 95% CI 2-sided [-8.8 to -5.5]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.2, 95% CI 2-sided [-10.9 to -7.5]

4. Secondary Outcome: Percentage of Participants Who Achieve ≥10% Body Weight Reduction
Description: Percentage of Participants who Achieve ≥10% Body Weight Reduction. A logistic regression model was used for this analysis.
Time Frame: Week 52
Population: All participants who received at least one dose of study drug and had evaluable body weight data.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
Percentage of participants | 70.0 | 83.82 | 14.71
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.19, 95% CI 2-sided [5.63 to 30.89]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.58, 95% CI 2-sided [11.23 to 72.71]

5. Secondary Outcome: Percentage of Participants Who Achieve ≥15% Body Weight Reduction
Description: Percentage of Participants who Achieve ≥15% Body Weight Reduction. A logistic regression model was used for this analysis.
Time Frame: Week 52
Population: All participants who received at least one dose of study drug and evaluable body weight data.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
Percentage of participants | 48.57 | 72.06 | 2.94
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 25.64, 95% CI 2-sided [6.68 to 98.49]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 69.79, 95% CI 2-sided [17.69 to 275.37]

6. Secondary Outcome: Mean Change From Baseline in Waist Circumference
Description: Mean Change from Baseline in Waist Circumference. LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable waist circumference data.
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
centimeters (cm) | -11.9 (0.83) | -16.4 (0.85) | -2.7 (0.84)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.2, 95% CI 2-sided [-11.5 to -6.9]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.7, 95% CI 2-sided [-16.0 to -11.3]

7. Secondary Outcome: Mean Change From Baseline in Absolute Body Weight
Description: Mean Change from Baseline in Absolute Body Weight. LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
kilograms (kg) | -13.1 (0.93) | -18.1 (0.95) | -2.1 (0.94)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -10.9, 95% CI 2-sided [-13.5 to -8.3]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -16.0, 95% CI 2-sided [-18.6 to -13.4]

8. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI)
Description: Mean Change from Baseline in BMI. LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable BMI data.
Measure: Least Squares Mean (Standard Error); unit: kilograms per metres squared (kg/m^2)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 70 | 68 | 68
kilograms per metres squared (kg/m^2) | -4.7 (0.29) | -6.4 (0.30) | -0.8 (0.30)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -3.9, 95% CI 2-sided [-4.8 to -3.1]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -5.6, 95% CI 2-sided [-6.4 to -4.8]

9. Secondary Outcome: Mean Change From Baseline in Hemoglobin A1c (HbA1c)
Description: Mean Change from Baseline in HbA1c. LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: all participants who received at least one dose of study drug and had evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 69 | 66 | 67
Percentage of HbA1c | -0.34 (0.032) | -0.35 (0.033) | 0.03 (0.033)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.37, 95% CI 2-sided [-0.46 to -0.28]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.39, 95% CI 2-sided [-0.48 to -0.29]

10. Secondary Outcome: Mean Change From Baseline in Fasting Glucose (FSG)
Description: Mean Change from Baseline in FSG. LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable fasting glucose data.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 69 | 66 | 67
millimoles per liter (mmol/L) | -0.25 (0.050) | -0.33 (0.052) | 0.22 (0.051)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.46, 95% CI 2-sided [-0.61 to -0.32]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.54, 95% CI 2-sided [-0.69 to -0.40]

11. Secondary Outcome: Mean Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score
Description: The SF-36v2 acute form, 1-week recall assesses participants' health-related quality of life (HRQoL) on 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Information from these 8 domains is further aggregated into 2 health component summary scores: Physical Component Summary and Mental Component Summary.
  Items are answered on Likert scales of varying lengths. Scoring of each domain and both summary scores are norm based and presented in the form of T scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function and/or better health. Range cannot be specified in norm-based scores.
  LS mean was determined using analysis of covariance (ANCOVA) model using Baseline + Sex + Presence of comorbidities + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable SF-36v2 data.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 58 | 58
Score on a scale | 2.0 (0.40) | 1.9 (0.42) | 0.8 (0.41)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.044, ANCOVA; LS Mean Difference = 1.2, 95% CI 2-sided [0.0 to 2.3]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.050, ANCOVA; LS Mean Difference = 1.2, 95% CI 2-sided [0.0 to 2.3]

12. Secondary Outcome: Mean Change From Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score
Description: The IWQOL Lite-CT consists of 20 items, assessing 2 primary domains of obesity related HRQoL: Physical (7 items) and Psychosocial (13 items). A 5-item subset of the Physical domain - the Physical Function composite - is also supported. Items in the Physical Function composite describe physical impacts related to general and specific physical activities. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better quality of life. LS mean was determined using ANCOVA model with Baseline + Sex + Presence of comorbidities + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable IWQOL-Lite-CT data.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 62 | 58 | 58
Score on a scale | 11.2 (1.44) | 12.0 (1.48) | 3.5 (1.48)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 7.8, 95% CI 2-sided [3.7 to 11.8]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 8.5, 95% CI 2-sided [4.4 to 12.7]

13. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (DBP) (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: LS mean was determined using MMRM model with Variable = Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury (mmHg)
Groups:
- Tirzepatide Pooled Analysis: Participants of 10 mg and 15 mg tirzepatide arms were pooled in this arm.
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 119 | 58
millimeters of Mercury (mmHg) | -6.1 (0.62) | -1.3 (0.88)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -4.8, 95% CI 2-sided [-6.9 to -2.7]

14. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: LS mean was determined using MMRM model with Baseline + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury (mmHg)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 119 | 58
millimeters of Mercury (mmHg) | -9.6 (0.87) | -3.5 (1.24)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.1, 95% CI 2-sided [-9.1 to -3.1]

15. Secondary Outcome: Mean Change From Baseline in Total Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: LS mean was determined using MMRM model using log (Actual measurement/Baseline) = log (Baseline) + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 123 | 61
millimoles per liter (mmol/L) | -0.37 (0.055) | -0.06 (0.085)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = -0.31, 95% CI 2-sided [-0.51 to -0.11]

16. Secondary Outcome: Mean Change From Baseline in High Density Lipoprotein (HDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: LS mean was determined using MMRM model using log (Actual Measurement) = log (Baseline) + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 123 | 61
millimoles per liter (mmol/L) | 0.12 (0.017) | 0.03 (0.023)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = 0.09, 95% CI 2-sided [0.03 to 0.14]

17. Secondary Outcome: Mean Change From Baseline in Low Density Lipoprotein (LDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: as for outcome 14
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 123 | 61
millimoles per liter (mmol/L) | -0.17 (0.056) | -0.11 (0.081)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = -0.06, 95% CI 2-sided [-0.25 to 0.13]

18. Secondary Outcome: Mean Change From Baseline in Very Low Density Lipoprotein (VLDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: as for outcome 16
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 123 | 61
millimoles per liter (mmol/L) | -0.28 (0.019) | -0.03 (0.042)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = -0.25, 95% CI 2-sided [-0.34 to -0.16]

19. Secondary Outcome: Mean Change From Baseline in Triglycerides (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: as for outcome 16
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 123 | 61
millimoles per liter (mmol/L) | -0.63 (0.045) | -0.05 (0.099)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = -0.58, 95% CI 2-sided [-0.79 to -0.37]

20. Secondary Outcome: Mean Change From Baseline in Free Fatty Acids (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: as for outcome 16
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 123 | 61
millimoles per liter (mmol/L) | -0.16 (0.013) | -0.10 (0.023)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = -0.07, 95% CI 2-sided [-0.12 to -0.01]

21. Secondary Outcome: Mean Change From Baseline in Fasting Insulin (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: LS mean was determined using MMRM model with log (Actual Measurement) = log (Baseline) + Sex + Presence of comorbidities + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable fasting insulin data.
Measure: Least Squares Mean (Standard Error); unit: milliunits per liter (mU/L)
Arm/Group | Tirzepatide Pooled Analysis | Placebo
Number analyzed (Participants) | 135 | 66
milliunits per liter (mU/L) | -6.5 (0.42) | -0.2 (1.09)
Statistical Analysis 1: Comparison: Tirzepatide Pooled Analysis vs Placebo; Test type: Superiority; LS Mean Difference = -6.3, 95% CI 2-sided [-8.6 to -4.0]

ADVERSE EVENTS:
Time Frame: Baseline Through Safety Follow-Up (Up To Week 56)
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Per protocol, adverse event analysis was planned as per the treatment regimen received.
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71 | 0/69
Serious Adverse Events (participants affected / at risk) | 3/70 | 8/71 | 6/69
Other Adverse Events (participants affected / at risk) | 61/70 | 56/71 | 39/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg Tirzepatide (N=70) | 15 mg Tirzepatide (N=71) | Placebo (N=69)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0/35 (0) | 0/36 (0) | 1/36 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1/35 (1) | 0/35 (0) | 0/33 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0/35 (0) | 0/35 (0) | 1/33 (1)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg Tirzepatide (N=70) | 15 mg Tirzepatide (N=71) | Placebo (N=69)
Abdominal distension (Gastrointestinal disorders) | 13 (62) | 9 (40) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (10) | 2 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 28 (121) | 29 (109) | 6 (11)
Flatulence (Gastrointestinal disorders) | 6 (13) | 6 (13) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (57) | 23 (79) | 4 (11)
Vomiting (Gastrointestinal disorders) | 8 (23) | 14 (53) | 3 (3)
Injection site reaction (General disorders) | 4 (11) | 2 (6) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (4) | 1 (2) | 6 (7)
Gastroenteritis (Infections and infestations) | 8 (9) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (25) | 17 (20) | 12 (13)
Vaginal infection (Infections and infestations) | 1/35 (1) | 2/35 (2) | 3/33 (3)
Amylase increased (Investigations) | 5 (5) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 5 (6) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 19 (75) | 20 (72) | 8 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 8 (8)
Dizziness (Nervous system disorders) | 2 (2) | 4 (37) | 3 (3)
Menstruation irregular (Reproductive system and breast disorders) | 2/35 (2) | 0/35 (0) | 1/33 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6) | 0 (0)
Abortion induced (Surgical and medical procedures) | 3/35 (3) | 1/35 (1) | 1/33 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT05024032/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT05024032/SAP_001.pdf